CLINICAL TRIAL: NCT01270932
Title: An Open-label, Pharmacokinetic Study of Lenalidomide (Revlimid) and High-dose Dexamethasone Induction Therapy in Previously Untreated Multiple Myeloma Patients With Various Degrees of Renal Dysfunction - Validation of Official Dosing Guidelines for Renal Failure
Brief Title: Lenalidomide & High Dose Dexamethasone for Untreated Multiple Myeloma Renal Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-PI-0505
Record Dates: First submitted 2010-12-13; First posted 2011-01-05 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Renal Failure; Multiple Myeloma
MeSH Terms: conditions — Renal Insufficiency; Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide and Dexamethasone (Experimental): Lenalidomide:Daily for 21 days of a 28 day cycle
  Dexamethasone:Days 1-4, 9-12, 17-20 for the first cycle and then weekly dexamethasone from cycles 2-4.
  Interventions: Drug: Lenalidomide and Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide and Dexamethasone — Lenalidomide:Daily for 21 days of a 28 day cycle Dexamethasone:Days 1-4, 9-12, 17-20 for the first cycle and then weekly dexamethasone from cycles 2-4.
  Other Names: Revlimid for Lenalidomide; Decadron for Dexamethasone

SUMMARY:
Primary:

• To validate the initial dosing recommendations for newly diagnosed MM (Mutiple Myeloma) patients with various degrees of renal failure using pharmacokinetic studies

Secondary:

* To evaluate the safety of lenalidomide and dexamethasone as induction therapy in newly-diagnosed MM (Multiple Myeloma) patients with renal dysfunction using modified dosing guidelines
* To evaluate clinical response of lenalidomide and dexamethasone after 4 cycles using the modified dosing guidelines
* To evaluate the ability to collect stem cells after 4 cycles of lenalidomide and dexamethasone induction therapy in MM (Multiple Myeloma) patients with renal failure

DETAILED DESCRIPTION:
STUDY DESIGN:

This is a single institution open label, pharmacokinetic validation study of the combination of lenalidomide with dexamethasone for firstline induction therapy in transplant-eligible MM ( Multiple Myeloma ) patients with various degrees of renal failure. There will be 4 patient groups with various degrees of renal function (based on creatinine clearance calculated from a 24 hour urine collection and requirement for dialysis). Each group will receive lenalidomide dosing as per official recommended guidelines:

Group 1 Normal {CrCl(creatinine clearance)>60 mL/min}25 mg (full-dose)-Daily for 21 days of a 28 Day cycle1 Group 2 Moderate renal impairment {30 ≤ CrCl (creatinine clearance) <60 mL/min}10 mg Daily for 21 days of a 28 day cycle Group 3 Severe renal impairment {CrCl (creatinine clearance)<30 mL/min, not requiring dialysis}15 mg Every 48 hours for 21 days of a 28 day cycle (11 PLANNED DOSES EACH 28 DAY CYCLE) Group 4 End-stage renal failure {CrCl (creatinine clearance)<30 mL/min, requiring dialysis}5 mg Once daily for 21 days of a 28 day cycle On dialysis days the dose should be administered following dialysis.

Pharmacokinetic (PK) studies: We will be evaluating PK studies following single and multiple doses of lenalidomide during Cycle 1.Patients will receive their first dose of lenalidomide (Cycle 1, day 1) as per the above designated patient group. PK (pharmacokinetic)sampling for 1st dose only will be drawn at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours post-dose for group 1 and at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48, 72 hours for all other groups. The 2nd dose of lenalidomide will be administered on Day 4 for all patients (i.e. no doses on Days 2 and 3). On Day 17 (after 14 doses of lenalidomide administered), repeat PK sampling will be performed at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours for groups 1, 2 and 4 (before next hemodialysis for those in group 4). Repeat PK sampling for group 3 will be performed at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following inclusion/exclusion criteria to be eligible for the study.

Inclusion criteria

Patients must fulfill all of the following criteria to be eligible for admission to the study:

1. Understand and voluntarily sign an informed consent form
2. Age≥18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Previously untreated, symptomatic multiple myeloma as defined by ALL 3 criteria below:

   * Monoclonal plasma cells in the bone marrow ≥10% and/or presence of a biopsy-proven plasmacytoma
   * Monoclonal protein present in the serum and/or urine
   * Myeloma-related organ dysfunction (at least one of the following):

   C - Calcium elevation in blood (serum calcium >upper limit of normal) R - Renal insufficiency (serum creatinine >177umol/L) A - Anemia (hemoglobin <100g/L or 20g/L below normal) B - Lytic bone lesions or osteoporosis
5. Eligible for autologous stem cell transplantation as per Princess Margaret Hospital criteria.
6. Disease measurable by serum or urine M (monoclonal) protein, free light chain assay, bone marrow plasmacytosis or plasmacytoma.
7. No prior myeloma therapy (Exception: up to 480 mg of dexamethasone is allowed within the past 28 days, as well as palliative, localized radiation therapy, without the requirement of a washout period prior enrollment).
8. ECOG (Eastern Cooperative Oncology Group) performance status of ≤ 2 at study entry.
9. Laboratory test results within these ranges:

   * Absolute neutrophil count ≥ 1,000/mm³
   * Platelet count ≥ 50,000/mm³ (untransfused)
   * Total bilirubin ≤ 22 umol/L
   * Aspartate transaminase (AST) also called serum glutamic oxaloacetic transaminase (SGOT) and Alanine transaminase (ALT) also called serum glutamic pyruvic transaminase (SGPT) ≤ 2 x ULN (upper limit number) or ≤ 5 x ULN if hepatic metastases are present.
   * Renal function must be measured by 24hour urine for creatinine clearance (CrCl) - any level of CrCl is allowed for eligibility.
10. Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
11. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL ( milli-International Units per milliliter ) within 7 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP (Females of childbearing potential) must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
12. Able to take aspirin 81mg daily as prophylactic anticoagulation [patients intolerant to ASA (Acetyl Salicylic acid - Aspirin) may use low molecular weight heparin].

Exclusion Criteria:

* Patients who fulfill any of the following criteria are not eligible for admission to the study:

  1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
  2. Pregnant or breast-feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
  3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
  4. Use of any other experimental drug or therapy, except for up to 480 mg of dexamethasone or palliative, localized radiation therapy, without the requirement of a washout period prior enrollment.
  5. Known hypersensitivity to thalidomide.
  6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
  7. Any prior use of lenalidomide.
  8. Concurrent use of other anti-cancer agents or treatments.
  9. Known positive for HIV (Human immunodeficiency virus) or infectious hepatitis, type B or C.
  10. Evidence of AL (amyloid light chain) amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-11; Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Serum Pharmacokinetic (PK) analysis of Study drug Lenalidomide | 16 months
  PK data will be analyzed and reported after completion of PK studies in all patients

SECONDARY OUTCOMES:
Evaluable for toxicity | 5 months
  All patients will be evaluable for toxicity from the time of their first treatment with Lenalidomide and dexamethasone.
Evaluable for response | 5 months
  All patients who have received at least 1 cycle of therapy and have their disease re-evaluated will be considered evaluable for response.
Overall and progression free survival rates which will be calculated by the method of Kaplan and Meier. | 16 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network- Princess Margaret Hosptial, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chen CI, Cao Y, Trudel S, Reece DE, Kukreti V, Tiedemann R, Prica A, Paul H, Le LW, Levina O, Kakar S, Lau A, Chen H, Chen E. An open-label, pharmacokinetic study of lenalidomide and dexamethasone therapy in previously untreated multiple myeloma (MM) patients with various degrees of renal impairment - validation of official dosing guidelines. Leuk Lymphoma. 2020 Aug;61(8):1860-1868. doi: 10.1080/10428194.2020.1747064. Epub 2020 May 31. PMID 32476520